CLINICAL TRIAL: NCT04294134
Title: MIO-CPP to Improve the Well-being, Permanency, and Safety Outcomes for Young Children at Risk of or in Out-of-home Placement in Philadelphia and Bucks Counties, and Affected by Pre and Post-natal Maternal Substance Use
Brief Title: MIO-CPP to Improve the Well-being, Permanency, and Safety Outcomes for Young Children at Risk of or in Out-of-home Placement in Philadelphia and Bucks Counties, and Affected by Maternal Substance Use
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Health Federation of Philadelphia (Other); Libertae, Inc. (Unknown); Gaudenzia Hutchinson Place (Unknown); Gaudenzia Winner Program (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-015904
Record Dates: First submitted 2020-02-21; First posted 2020-03-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Substance Use Disorders; Parent-Child Relations; Parent Child Abuse
Keywords: Child-parent therapy; Reflective parenting; Trauma-informed care
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: We will use a quasi-experimental trial design with historical controls as well as qualitative interviews to assess effectiveness and efficiency of MIO-CPP when paired with CRS, on parent and child outcomes including therapy engagement, parent/caregiver well-being, child well-being, and family well-being. The study will take place over two phases. Eligible caregivers in Phase 1 will receive MIO-CPP (control), while participants enrolled in Phase 2 will receive a MIO-CPP while also being paired with a CRS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIO-CPP (Active Comparator): The 9 month MIO-CPP model will begin with the standard 12 weeks of MIO for each mother, with the CPP assessment and engagement phase embedded during this time. This phase will be followed by the dyadic mother-child phase, the core intervention stage of CPP. If a parent needs additional stabilization, more individual time can be added. During the core phase of dyadic CPP the Child Parent Specialists will continue to build and strengthen parents' reflective functioning by embedding aspects from MIO. The 9 month MIO-CPP model will begin with the standard 12 weeks of MIO for each mother, with the CPP assessment and engagement phase embedded during this time. This phase will be followed by the dyadic mother-child phase, the core intervention stage of CPP. If a parent needs additional stabilization, more individual time can be added.
  Interventions: Behavioral: MIO-CPP
- MIO-CPP-CRS (Experimental): In Phase 2, participants will receive MIO-CPP therapy, as well as support from a CRS. The MIO-CPP model will begin with 6 sessions of MIO for each study participant, with the CPP assessment and engagement phase embedded during this time. This phase will be followed by the dyadic mother-child phase, the core intervention stage of CPP. If a parent needs additional stabilization, more individual time can be added. During the core phase of dyadic CPP the Child Parent Specialists will continue to build and strengthen parents' reflective functioning by embedding aspects from MIO.
  Participant dyads will be assigned a Certified Recovery Specialists (CRSs) who will provide services to support them as they transition out of SUD treatment and back into their home communities.
  Interventions: Behavioral: MIO-CPP-CRS

INTERVENTIONS:
Behavioral: MIO-CPP — Mothering from the Inside Out (MIO) is an individual, 12-session, manualized, psychotherapeutic intervention designed to promote parental reflective functioning in mothers who are in treatment for SUDs and/or other mental health problems, and caring for a child in-utero through five years old. (Suchman N, Pajulo M, and Mayes LC, 2013).
  Child-Parent Psychotherapy (CPP) is a two-generation approach that supports and strengthens parent-child attachment by integrating modalities derived from psychodynamic, attachment, trauma, cognitive-behavioral, and social learning theories. (Lieberman AF and Van Horn P, 2005 and 2008) Studies have revealed that CPP caregivers' outcomes include decreased depression, PTSD and other symptoms, increased empathy towards children and an increase in the quality of parent-child interactions. CPP focuses on working with families offering weekly sessions for nine-12 months.
  Arms: MIO-CPP
Behavioral: MIO-CPP-CRS — Mothering from the Inside Out (MIO) is an individual, 12-session, manualized, psychotherapeutic intervention designed to promote parental reflective functioning in mothers who are in treatment for SUDs and/or other mental health problems, and caring for a child in-utero through five years old. (Suchman N, Pajulo M, and Mayes LC, 2013).
  Child-Parent Psychotherapy (CPP) is a two-generation approach that supports and strengthens parent-child attachment by integrating modalities derived from psychodynamic, attachment, trauma, cognitive-behavioral, and social learning theories. (Lieberman AF and Van Horn P, 2005 and 2008) CPP focuses on working with families offering weekly sessions for nine-12 months.
  Certified Recovery Specialists (CRS) provide peer support services are an evidence-based…model of care which consists of a qualified peer support provider who assists individuals with their recovery from mental illness and substance use disorders.
  Arms: MIO-CPP-CRS

SUMMARY:
The goal of the project is to improve child well-being, permanency, and safety, and reduce the risk for involvement in the child welfare system for families with children pre-birth to five years who are affected by parental substance use disorders (SUD). The project will integrate with SUD treatment programs for pregnant/parenting women and their children and provide an evidence-based therapeutic model, Mothering from the Inside Out (MIO) and Child Parent Psychotherapy (CPP). MIO-CPP promotes the development of parental reflective functioning and strengthen parent/child attachment. The project will also examine the role of Certified Recovery Specialists (CRS) to provide case management services to parents during their enrollment in therapy.

MIO is an individual, manualized, psychotherapeutic intervention designed to promote parental reflective functioning in mothers who are in treatment for SUDs and/or other mental health problems, and caring for a child in-utero through five years old. CPP is typically offered through weekly sessions with the mother-child dyad that last 1 to 1.5 hours.

The MIO-CPP (intervention) model will begin with 6 sessions of MIO for each study participant, with the CPP assessment and engagement phase embedded during this time. This phase will be followed by the dyadic mother-child phase, the core intervention stage of CPP. If a parent needs additional stabilization, more individual time can be added. During the core phase of dyadic CPP the Child Parent Specialists will continue to build and strengthen parents' reflective functioning by embedding aspects from MIO.

Beginning in Phase 2, participant dyads will be assigned a Certified Recovery Specialists (CRSs) who will provide services to support them as they transition out of SUD treatment and back into their home communities. We will recruit and hire 2 PA CRSs to join the therapeutic team. CRS services will include but not be limited to: assisting clients with securing housing and employment and connecting to outpatient and other recovery support services (e.g. 12-step programs), and child, medical and behavioral health care as needed. The plan for the timing to introduce CRS services and their issues of focus will be defined through quality improvement methodology during Phase 1.

We will use a quasi-experimental trial design with historical controls as well as qualitative interviews to assess effectiveness and efficiency of MIO-CPP when paired with CRS, on parent and child outcomes including therapy engagement, parent/caregiver well-being, child well-being, and family well-being. The study will take place over two phases. Eligible caregivers in Phase 1 will receive MIO-CPP (control), while participants enrolled in Phase 2 will receive a MIO-CPP while also being paired with a CRS.

The recruitment for study participants will stop when 320 mother-child dyads have enrolled in the study. Participants will include mother-child dyads from families involved with residential SUD treatment programs serving women and children in Philadelphia and Bucks counties. In Bucks County we will receive referrals from Libertae Inc. in Bensalem, Pennsylvania (PA). In Philadelphia, we will receive referrals from Gaudenzia Hutchinson Place and the Gaudenzia Winner Program.

Data collection from participants will occur at four time points during the study: 1) when participants are enrolled; 2) 3 months following enrollment; 3) 6 months following enrollment; and 4) 9 months following enrollment or when the participant ends their participation in weekly therapy sessions if sooner than 9 months following enrollment. Study measures will include: 1) Parent/Caregiver Well-being: a) maternal reflective functioning, b) depression, anxiety, and trauma-related symptoms, c) parental substance use and move toward recovery; d) parenting stress; e) parent-child relationship; 2) Child Well-being: a) behavior problems, b) executive functions; c) socialization skills; 3) Family Well-being: a) child welfare involvement, b) reunifications.

As part of this study, investigator will acquire administrative data about the safety and permanency of children and adult recovery for all study participants. The Primary Investigator will request substance use treatment data from the City of Philadelphia Department of Human Services. The requested data elements will include whether the study child has a child welfare record, the types of allegations of abuse or neglect, and when the allegations occurred (from birth to present day). Additionally, investigators will request all available substance use treatment records will be requested for adults who are a part of a study case for the year prior to enrollment in the study to one year following their enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Women actively receiving treatment for Substance Use Disorder at one of three participating residential substance use disorder clinics in Philadelphia and Bucks Counties (Libertae Inc.; Gaudenzia's Hutchinson House; Gaudenzia Winner Program).
2. Must be at least six months pregnant or must have a child 5 years old or younger.
3. Must have access to child - children must either reside with mother, or, if the child is in foster/kinship care, the goal must be reunification.

Exclusion Criteria:

1. Duration of affiliation with treatment center:

   Women will not be referred for enrollment before they have been affiliated with the treatment facility for at least 14 days and will not be referred if they are less than 45 days from discharge.

   These limitations will ensure that women are not referred to our study too quickly as they are adjusting to residential treatment, but will also ensure that we do not enroll women too soon before they are discharged from residential treatment.
2. Non-English Speaking The study will not enroll mothers who would be unable to receive the intervention services in English without the assistance of an interpreter. Due to the duration of the study intervention as well as the frequency of visits between the Child-Parent Specialist and the client, it would not be feasible to ensure that an interpreter would also be available for all visits.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Infant/Toddler Sensory Profile (ITSP) | Baseline and 9 months
  The ITSP provides a standard method for professionals to measure a child's sensory processing abilities and to profile the effect of sensory processing on functional performance in the daily life of a child. This instrument is required as part of the cross-site evaluation.
  The ITSP is a judgment-based caregiver questionnaire. Each item describes children's responses to various sensory experiences. The ITSP consists of 36 items for children - birth to 6 months - and 48 items for children - 7 to 36 months. The questionnaire is available in English and Spanish. The caregiver questionnaire contains items divided into sensory systems. For children birth to 6 months, there are four quadrant scores and one combined quadrant score; for children 7 to 36 months, there are five sensory processing section scores, four quadrant scores, and one combined quadrant score available.
Change in Infant Traumatic Stress Questionnaire (ITSQ) | Baseline and 9 months
  The ITSQ is an 18-item questionnaire based on 3 of the 4 general criteria for diagnosis of Traumatic Stress Disorder in the Diagnostic Classification: 0-3. The ITSQ is used with children under two. For each tool, the three general criteria sampled were "numbing," "increased arousal," and "fears or aggression." The instruments are completed by parents. The participant responds "Yes" or "No" to each question and scores are summed.
Change in Child Traumatic Stress Questionnaire (CTSQ) | Baseline and 9 months
  The CTSQ is a 27-item questionnaire based on the criteria for the diagnosis of Traumatic Stress Disorder in the Diagnostic and Statistical Manual of Mental disorders research scale (DSM-IV-RS) and the DC: 0 - 3. The CTSQ with children ages 2 through 4. For each tool, the three general criteria sampled were "numbing," "increased arousal," and "fears or aggression." The instruments are completed by parents. The participant responds "Yes" or "No" to each question and scores are summed.
Change in PSI-SF | Baseline and 9 months
  The Parenting Stress Index Short Form (PSI-short form), a 36-item symptom inventory designed to identify parent-child dyads experiencing stress and at risk for dysfunctional parenting and behavior problems. It uses 3 categories: parental distress, parent-child dysfunctional interaction, and difficult child.

SECONDARY OUTCOMES:
Adult-Adolescent Parenting Inventory (AAPI) | Baseline and 9 months
  The AAPI is an inventory designed to assess the parenting and child rearing attitudes of adolescents and adult parent and pre-parent populations. Based on the known parenting and child rearing behaviors of abusive parents, responses to the inventory provide an index of risk for practicing behaviors known to be attributable to child abuse and neglect. The AAPI-2.1 is the revised and re-normed version of the original AAPI. The AAPI-2 consists of Form A (administered at Baseline) and Form B (Administered at study exit).
Trauma Symptoms Checklist (TSC-40) | Baseline and 9 months
  The TSC-40 is a 40-item self-report measure of symptomatic distress in adults arising from childhood or adult traumatic experiences. It measures aspects of posttraumatic stress as well as other symptoms found in some traumatized individuals.
  Respondents are asked to rate how often they have experienced each symptom in the last two months using a 4-point frequency rating scale ranging from 0 ("never") to 3 ("often"). In addition to yielding a total score (ranging from 0 to 120), the TSC-40 has six subscales: Anxiety, Depression, Dissociation, Sexual Abuse Trauma Index, Sexual Problems, and Sleep Disturbances.
Addiction Severity Index (ASI) | Baseline and 9 months
  The ASI is a semi-structured interview designed to address seven potential problem areas in substance-abusing patients: medical status, employment and support, drug use, alcohol use, legal status, family/social status, and psychiatric status. In 1 hour, a skilled interviewer can gather information on recent (past 30 days) and lifetime problems in all of the problem areas. The ASI provides an overview of problems related to substance, rather than focusing on any single area.
Child Behavior Checklist (CBCL) | Baseline and 9 months
  The Child Behavior Checklist is part of the Achenbach System of Empirically Based Assessment (ASEBA) and use information collected from parents to assess the behavior and emotional and social functioning of children. For this project, we will be using the Preschool Form, which is appropriate for children ages 18 to 71 months (5 years). Primary caregivers rate their children for how true each item is now or in the past six months as not true, somewhat or sometimes true, or very true or often true. The form takes approximately 10 to 15 minutes to complete. The 99 items in the preschool CBCL are organized into two broad groupings of seven syndromes.
Center for Epidemiologic Studies - Depression Scale Short Form (CESD-SF) | Baseline, 3 months, 6 months, and 9 months
  The CES-D-SF is a screening tool used to assess the presence and severity of depressive symptoms occurring over the past week. The CES-D-SF measures four factors related to depression: depressive affect, somatic symptoms, positive affect, and interpersonal relations. Total scores are calculated, which can be used to classify people as having little/no risk of depression, mild to moderate depression, or possibly severe depression. The short form of this self-administered questionnaire takes fewer than 10 minutes to complete. The CES-D-SF may be self or interviewer-administered.
PC-PTSD-5 | Baseline, 3 months, 6 months, and 9 months
  The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) is a 5-item screen that was designed for use in primary care settings. The measure begins with an item designed to assess whether the respondent has had any exposure to traumatic events. If a respondent denies exposure, the PC-PTSD-5 is complete with a score of 0. However, if a respondent indicates that they have experienced a traumatic event over the course of their life, the respondent is instructed to respond to five additional yes/no questions about how that trauma exposure has affected them over the past month. The PC-PTSD-5 was designed to identify respondents with probable PTSD.
Keys to Interactive Parenting (KIPS) | Baseline, 3 months, 6 months, and 9 months
  The quality of parent-child interactions will measured by video recording each selected parent (of the subset) interacting with his/her child for 20 minutes and then analyzing the video data using The Keys to Interactive Parenting Scale (KIPS). KIPS is a structured observation tool of parent-child interaction. It uses play time to assess 12 parenting behaviors.
Parenting Relationship Questionnaire (PRQ) | Baseline and 9 months
  The Parenting Relationship Questionnaire (PRQ) is designed to capture a parent's perspective on the parent-child relationship. The PRQ has two forms, one for parents of preschool children (aged 2-5) and one for parents of children and adolescents (age 6-18). We will use the preschool version of the assessment, which can be completed in 10-15 minutes. The PRQ (Parenting Relationship Questionnaire) instrument is designed to capture a parent's perspective of the parent-child relationship (or the perspective of a person serving a similar role). It assesses traditional parent-child dimensions such as attachment and involvement and also provides information on parenting style, parenting confidence, stress, and satisfaction with the child's school. The questionnaire is designed to be used in clinical, pediatric, counseling, school, and other settings where there is a need to understand the nature of the parent-child relationship.
Parent Development Interview (PDI) | Baseline and 9 months
  The PDI is a 45 item video-taped, semi-structured clinical interview intended to examine parents' representations of their children, themselves as parents, and their relationships with their children. The PDI is intended to assess internal working models of relationships. The PDI elicits representations regarding a current, ongoing, "live" relationship that is still evolving, that of the parent with her or his child. The parent is asked to describe her or his child's behavior, thoughts, and feelings in various situations, as well as her responses to her or his child in these situations. The parent is also asked to describe him/herself as a parent and to discuss emotions stimulated by the experience of parenting. The interview strives in a number of ways to tap into parents' understanding of their child's behavior, thoughts, and feelings, and asks the parents to provide real life examples of charged interpersonal moments: "Describe a time in the last week when you and your child really
Pregnancy Interview | Baseline
  Like the Parent Development Interview (PDI), the Pregnancy Interview (PI) is a 45-minute semi-structured video-taped, semi-structured clinical interview that has been shown to predict to adult attachment classification. It has 39 questions and probes and was developed to assess the quality of a mother's representation of her relationship with her unborn child. The interview, which is administered during the third trimester, assesses a variety of aspects of the mother's view of her emotional experience with pregnancy and her expectations and fantasies regarding her future relationship with her child.
  The PI is only used at Baseline because it can only be administered to people who are currently pregnant. Baseline is the only time point when a participant would be currently pregnant. For women who complete the pregnancy interview at Baseline, they would instead complete the PDI at Program Exit.

OTHER OUTCOMES:
Child welfare involvement | On year prior to study enrollment and one year following study exit
  Safety and permanency records for the child will be requested (from birth to one year following study exit) for children who are a part of the study case. Records will be obtained by providing the appropriate agency with the necessary identifying information (name, date of birth, and social security number) needed to identify the requested records. These records will be obtained for the period 12 months prior to study enrollment until 12 months following exit from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Matone, DrPH, MHS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Roberts Center for Pediatric Research, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
For all study participants, study staff are required to share the following data elements for each study participant with the Children's Bureau, Mathematica Policy Research Institute, and Walter R. McDonald & Associates (WMRA): 1) administrative data regarding safety and permanency records for the child (from birth to present day) for children who are a part of a study case; 2) substance use treatment records for adults (from age 18 to present day) who are a part of a study case from one year prior to study enrollment to one year following study exit; 3) all participant responses to study questionnaires; and 4) dates of enrollment, service logs and dates of service from each of the participant's encounters with a Child-Parent Specialist, and case closure; 5) child's date of birth. Data will be reported using the Department of Health and Human Services' secure web-based platform, RPG-EDS.
Time Frame: Deidentified participant data will be available following completion of all study activities for all grantees in the Children's Bureau Regional Partnership Grant (RPG7) in accordance with Child and Family Services Improvement and Innovation Act (Pub. L. 112 34) in order to evaluate grantee performance.
Access Criteria: Deidentified participant data will be shared with the Children's Bureau, Mathematica Policy Research Institute, and Walter R. McDonald & Associates (WMRA).

REFERENCES:
- [Background] Suchman N, Pajulo M, and Mayes LC, 2013. Parenting and Substance Abuse: Developmental Approaches and Interventions. "Mothering from the Inside Out: A Mentalization-Based Individual Therapy for Mothers with Substance-Use Disorders." Page 407. New York, NY: Oxford University Press.
- [Background] Lieberman, A. F., & Van Horn, P. (2005). Don't Hit My Mommy! A Manual for Child-Parent Psychotherapy With Young Witnesses of Family Violence. Washington, D.C. : Zero to Three Press.
- [Background] Lieberman, A. F., & Van Horn, P. (2008). Psychotherapy with Infants and Young Children: Repairing the Effects of Stress and Trauma on Early Attachment. New York: Guilford Press.